CLINICAL TRIAL: NCT04329338
Title: Effects of Lactobacillus Pentosus KCA1 on the Gut and Vaginal Microbiome of Women With Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nnamdi Azikiwe University (Other)
Responsible Party: Principal Investigator, Kingsley C Anukam, Reader/Research Scientist, Nnamdi Azikiwe University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NAUTH/CS/66/V046
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Bacterial Vaginoses
Keywords: Lactobacillus; Microbiota; Nigerian women; Gut; Vagina; 16S rRNA; Sequencing; Metagenomics
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: In this case each participant served as control as we collected sample before and after intervention
Masking Description: This is an open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gut and vaginal sample collection (No Intervention): Gut and vaginal samples were collected for Nugent score, and 16S rRNA metagenomics communities.
- Gut and Vaginal sample after Lactobacillus (Experimental): Seven women diagnosed with BV by Nugent score (7-10) provided vaginal and gut sample after 14 days oral intake of 3 grams (2.5X108 cfu/g) of Lactobacillus pentosus KCA1
  Interventions: Other: Lactobacillus pentosus KCA1

INTERVENTIONS:
Other: Lactobacillus pentosus KCA1 — Lactobacillus pentosus KCA1 suspended in dairy and taken orally for 14 days
  Arms: Gut and Vaginal sample after Lactobacillus

SUMMARY:
Bacterial vaginosis (BV) is under-reported, misdiagnosed and inappropriately treated in Nigeria. Treatment option rely on antibiotics that eliminates both good and pathogenic bacteria, with gross impact on the gut and vaginal microbiome. Our primary objective in this study is to determine the effects of Lactobacillus on the gut and vagina when taken orally.

DETAILED DESCRIPTION:
Antibiotics reduces in considerable proportion both the healthy bacteria especially Lactobacilli and those associated with BV, thus the vaginal microecology and gut is adversely affected. It is widely acknowledged that Lactobacilli and other genera that produces some metabolites such as lactic acid, contributes to vaginal health by maintaining the low pH of the vagina.

The objectives of this study are three folds, first to determine the effects before and after 14 days oral feeding of Lactobacillus pentosus KCA1 on the vaginal and gut microbiota compositions of women diagnosed with BV. Second to measure the level of two proinflammatory cytokines IL-1 beta and IL-6 before and after KCA1 consumption and third to determine in silico, the relative abundance of microbial genes involved in metabolic functions using the 16S rRNA datasets.

ELIGIBILITY:
Inclusion Criteria:

* Not on antibiotic therapy within the last one month
* Not menstruating at the time of inclusion.

Exclusion Criteria:

Pregnant, use of antibiotic medication, declined informed consent, menstruating and those that used douches, sprays, spermicides in the last 48 hours

-

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Nugent score | 14 days
  Gram stain microscopy for different bacterial morphotypes
Gut and Vaginal microbiota | 14 days
  Relative abundance of bacterial communities before and after Lactobacillus pentosus KCA1

SECONDARY OUTCOMES:
IL-6 Proinflammatory cytokine | 14 days
  Levels of Interleukin-6 with Enzyme-Linked Immunosorbent assay (ELISA)
IL-1beta Proinflammatory cytokine | 14 days
  Level of Interleukin-I beta with Enzyme-Linked Immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- Nnamdi Azikiwe University Teaching Hospital, Nnewi, Anambra, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anukam KC, Macklaim JM, Gloor GB, Reid G, Boekhorst J, Renckens B, van Hijum SA, Siezen RJ. Genome sequence of Lactobacillus pentosus KCA1: vaginal isolate from a healthy premenopausal woman. PLoS One. 2013;8(3):e59239. doi: 10.1371/journal.pone.0059239. Epub 2013 Mar 19. PMID 23527145